CLINICAL TRIAL: NCT03259789
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Bexagliflozin in Subjects With Type 2 Diabetes Mellitus Who Are Not Adequately Controlled by Metformin Alone
Brief Title: Safety and Efficacy of Bexagliflozin Compared to Placebo as Add-on Therapy to Metformin in Type 2 Diabetes Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THR-1442-C-419
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — bexagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bexagliflozin tablets, 20 mg; Double-Blind (Active Comparator)
  Interventions: Drug: Bexagliflozin tablets, 20 mg
- Bexagliflozin tablets, Placebo; Double Blind (Placebo Comparator)
  Interventions: Drug: Bexagliflozin tablets, placebo
- Bexagliflozin Tablets, 20 mg; High Glycemic Group (Experimental)
  Interventions: Drug: Bexagliflozin tablets, 20 mg

INTERVENTIONS:
Drug: Bexagliflozin tablets, 20 mg — Each subject will receive bexagliflozin, 20 mg once daily for the duration of the study.
  Other Names: EGT0001442, EGT0001474
  Arms: Bexagliflozin tablets, 20 mg; Double-Blind
Drug: Bexagliflozin tablets, placebo — Each subject will receive placebo (inactive tablet) once daily for the duration of the study.
  Arms: Bexagliflozin tablets, Placebo; Double Blind
Drug: Bexagliflozin tablets, 20 mg — Each subject will receive bexagliflozin, 20 mg once daily for the duration of the study.
  Other Names: EGT0001442, EGT0001474
  Arms: Bexagliflozin Tablets, 20 mg; High Glycemic Group

SUMMARY:
The purpose of this study is to investigate the effect of bexagliflozin compared to placebo as an add-on therapy to metformin in lowering hemoglobin A1c (HbA1c) levels in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Approximately 300 subjects with inadequately controlled T2DM on metformin were to be recruited from the United States and Japan. Subjects were randomly assigned to receive bexagliflozin tablets, 20 mg, or bexagliflozin tablets, placebo, in a ratio of 1:1 once daily for 24 weeks. Subjects were to continue taking metformin for the duration of the study. The study also enrolled 50 subjects with extremely poorly controlled T2DM on metformin to receive open-label bexagliflozin tablets, 20 mg, for 24 weeks.

ELIGIBILITY:
The subjects were required to meet the following criteria at the time of enrollment to be eligible for the study:

1. Had been age ≥ 20 years at screening. Women of childbearing potential were required to have tested negative for pregnancy and have agreed to abstinence or contraception for the duration of the study to avoid any possible pregnancy. Females who were surgically sterile (hysterectomy, oophorectomy) or postmenopausal (absence of menses greater than 12 months) were eligible if they had tested negative for pregnancy at screening.
2. a) Had a history of T2DM with an HbA1c level of ≥ 7.5% and ≤ 10.5% at screening, or b) Had a history of T2DM with an HbA1c level of >10.5% and ≤ 12.0% at screening
3. Had been prescribed a stable dose of metformin (≥1500 mg per day in the US or ≥ 1000 mg per day in Japan) as their sole anti-diabetic medication
4. Had a body mass index (BMI) ≤ 45 kg m-2
5. Had been able to comprehend and willing to provide written informed consent in accordance with institutional and regulatory guidelines
6. Had no recent changes to their medications for hypertension or hyperlipidemia (if applicable)
7. Had the ability to regularly self-administer medication, as evidenced by consumption of all, or at worst one less than all, doses of run-in medication prior to randomization

Subjects who met any of the following criteria were to be excluded from the study:

1. Had a diagnosis of type 1 diabetes mellitus or maturity-onset diabetes of the young
2. Were pregnant or breastfeeding
3. Had one or more hemoglobin alleles that affect HbA1c measurement
4. Had a history of genitourinary tract infection (e.g., UTI, GMI, vaginitis, balanitis) within 6 weeks of screening or a history of ≥ 3 genitourinary infections requiring treatment within 6 months of screening
5. Had an estimated glomerular filtration rate (eGFR), as calculated by the modification of diet in renal disease study equation (MDRD), < 60 mL min-1 per 1.73 m2
6. Had a sitting systolic blood pressure >180 mmHg or a sitting diastolic blood pressure > 110 mmHg at screening
7. Had exposure to hypoglycemic agent(s) other than metformin during the 8 weeks prior to screening
8. Had a history of illicit drug use or alcohol abuse in the past 2 years
9. Had a life expectancy < 2 years
10. Had a diagnosis of New York Heart Association (NYHA) Class IV heart failure within 3 months of screening
11. Had experienced an MI, unstable angina, stroke, or hospitalization for heart failure within 3 months of screening
12. Had exposure to an investigational drug within 30 days
13. Had a previous exposure to bexagliflozin or EGT0001474
14. Had a history of SGLT2 inhibitor treatment
15. Were participating in another interventional trial
16. Were not able to comply with the study scheduled visits
17. Had any condition, disease, disorder, or clinically relevant abnormality that, in the opinion of the primary investigator, would jeopardize the subject's appropriate participation in this study or obscure the effects of treatment
18. Had an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 × ULN or total bilirubin ≥ 1.5 × ULN at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J, Paul Lock, M.D., Study Director — Theracos
Locations (43):
- United States (26):
  - Clinical Research Site 1232, Birmingham, Alabama
  - Clinical Research Site 1378, Birmingham, Alabama
  - Clinical Research Site 1269, Foley, Alabama
  - Clinical Research Site 1363, Little Rock, Arkansas
  - Clinical Research Site 1381, Anaheim, California
  - Clinical Research Site 1375, North Hollywood, California
  - Clinical Research Site 1365, Norwalk, California
  - Clinical Research Site 1382, Norwalk, Connecticut
  - Clinical Research Site 1372, Hollywood, Florida
  - Clinical Research Site 1362, Palm Springs, Florida
  - Clinical Research Site 1373, Pembroke Pines, Florida
  - Clinical Research Site 1376, Nampa, Idaho
  - Clinical Research Site 1366, Chicago, Illinois
  - Clinical Research Site 1294, New Orleans, Louisiana
  - Clinical Research Site 1374, St Louis, Missouri
  - Clinical Research Site 1370, Las Vegas, Nevada
  - Clinical Research Site 1009, Berlin, New Jersey
  - Clinical Research Site 1037, Trenton, New Jersey
  - Clinical Research Site 1286, Albuquerque, New Mexico
  - Clinical Research Site 1368, New York, New York
  - Clinical Research Site 1275, The Bronx, New York
  - Clinical Research Site 1019, Portland, Oregon
  - Clinical Research Site 1379, Gonzales, Texas
  - Clinical Research Site 1369, Houston, Texas
  - Clinical Research Site 1371, San Antonio, Texas
  - Clinical Research Site 1360, San Antonio, Texas
- Japan (17):
  - Clinical Research Site 6048, Nagoya, Aichi-ken
  - Clinical Research Site 6050, Sapporo, Hokkaido
  - Clinical Research Site 6041, Koga, Ibaraki
  - Clinical Research Site 6029, Atsugi, Kanagawa
  - Clinical Research Site 6051, Kamakura, Kanagawa
  - Clinical Research Site 6020, Yokohama, Kanagawa
  - Clinical Research Site 6055, Tokyo, Meguro
  - Clinical Research Site 6046, Higashiosaka, Osaka
  - Clinical Research Site 6033, Kashihara, Osaka
  - Clinical Research Site 6013, Toyonaka, Osaka
  - Clinical Research Site 6052, Kawaguchi, Saitama
  - Clinical Research Site 6053, Shimotsuke, Tochigi
  - Clinical Research Site 6040, Fukuoka
  - Clinical Research Site 6043, Kyoto
  - Clinical Research Site 6015, Osaka
  - Clinical Research Site 6045, Tokyo
  - Clinical Research Site 6047, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-blind Group: Bexagliflozin 20 mg: Each subject will receive bexagliflozin, 20 mg, once daily and open-labeled metformin background medication during the entire study at a stable dose and frequency.
- Double-blind Group: Placebo: Each subject will receive placebo (inactive tablet) once daily and open-labeled metformin background medication during the entire study at a stable dose and frequency.
- High Glycemic Group: Each subject will receive Bexagliflozin tablet, 20 mg, once daily and open-labeled metformin background medication during the entire study at a stable dose and frequency.
Period: Overall Study
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo | High Glycemic Group
Started | 158 | 159 | 34
Completed | 141 | 142 | 28
Not Completed | 17 | 17 | 6
Not completed — Adverse Event | 3 | 2 | 1
Not completed — Withdrawal by Subject | 9 | 5 | 1
Not completed — Lost to Follow-up | 5 | 9 | 4
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Glycemic Group: Each subject will receive Bexagliflozin, 20 mg, once daily and open-labeled metformin background medication during the entire study at a stable dose and frequency.
- Total: Total of all reporting groups
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo | High Glycemic Group | Total
Number analyzed (Participants) | 158 | 159 | 34 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] — Total number of participants for Double-blind group is 317. The number of participants for High Glycemic group is 34. Population: For the Double-blind group, the High Glycemic group is excluded. Therefore, the number of participants analyzed is 317. Conversely, for the High Glycemic group, the Double-blind group is excluded. Therefore, the number of participants analyzed is 34.
  years
    Double-blind Group: number analyzed (Participants) | 158 | 159 | 0 | 317
    Double-blind Group | 56.0 (10.05) | 55.6 (11.18) |  | 55.8 (10.62)
    High Glycemic Group: number analyzed (Participants) | 0 | 0 | 34 | 34
    High Glycemic Group |  |  | 52.1 (8.59) | 52.1 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 65 | 15 | 138
  Male | 100 | 94 | 19 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 32 | 9 | 76
  Not Hispanic or Latino | 123 | 127 | 25 | 275
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 78 | 79 | 9 | 166
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 26 | 29 | 12 | 67
  White | 51 | 48 | 11 | 110
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 83 | 27 | 193
  Japan | 75 | 76 | 7 | 158
Height [Mean (Standard Deviation); unit: cm] — Total number of participants for Double-blind group is 317. The number of subjects for High Glycemic group is 34. Population: For the Double-blind group, the High Glycemic group is excluded. Therefore, the number of participants analyzed is 317. Conversely, for the High Glycemic group, the Double-blind group is excluded. Therefore, the number of participants analyzed is 34.
  cm
    Double-blind Group: number analyzed (Participants) | 158 | 159 | 0 | 317
    Double-blind Group | 168.4 (9.71) | 167.3 (9.55) |  | 167.8 (9.63)
    High Glycemic Group: number analyzed (Participants) | 0 | 0 | 34 | 34
    High Glycemic Group |  |  | 169.4 (9.34) | 169.4 (9.34)
Body Weight [Mean (Standard Deviation); unit: kg] — Total number of participants for Double-blind group is 317. The number of participants for High Glycemic group is 34. Population: For the Double-blind group, the High Glycemic group is excluded. Therefore, the number of participants analyzed is 317. Conversely, for the High Glycemic group, the Double-blind group is excluded. Therefore, the number of participants analyzed is 34.
  kg
    Double-blind Group: number analyzed (Participants) | 158 | 159 | 0 | 317
    Double-blind Group | 84.58 (21.989) | 84.44 (20.928) |  | 84.51 (21.43)
    High Glycemic Group: number analyzed (Participants) | 0 | 0 | 34 | 34
    High Glycemic Group |  |  | 87.28 (17.759) | 87.28 (17.759)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Total number of participants for Double-blind group is 317. The number of participants for High Glycemic group is 34. Population: For the Double-blind group, the High Glycemic group is excluded. Therefore, the number of participants analyzed is 317. Conversely, for the High Glycemic group, the Double-blind group is excluded. Therefore, the number of participants analyzed is 34.
  kg/m^2
    Double-blind Group: number analyzed (Participants) | 158 | 159 | 0 | 317
    Double-blind Group | 29.67 (6.45) | 29.99 (6.342) |  | 29.83 (6.388)
    High Glycemic Group: number analyzed (Participants) | 0 | 0 | 34 | 34
    High Glycemic Group |  |  | 30.37 (5.558) | 30.37 (5.558)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 24 for Double-blind Group
Description: HbA1c was obtained at baseline and at Week 24. The model-adjusted change from baseline was calculated using mixed-effects repeated measures analysis.
Time Frame: Baseline to week 24
Population: The intention-to-treat (ITT) population was used for the primary analysis. Subjects with a value at baseline and at week 24 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo
Number analyzed (Participants) | 142 | 145
percentage of HbA1c | -1.09 (0.076) | -0.56 (0.075)
Statistical Analysis 1: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures; Mixed-effects repeated measures analysis includes country, treatment, visit, treatment and baseline HbA1c value as fixed effect covariates; Difference of LS Means = -0.53, 95% CI 2-sided [-0.74 to -0.32]

2. Primary Outcome: Change From Baseline in HbA1c at Week 24 for High Glycemic Group
Description: The change in HbA1c from baseline at Week 24 in High Glycemic Group was calculated by subtracting the mean HbA1c at baseline from the mean HbA1c at Week 24
Time Frame: Baseline to week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | High Glycemic Group
Number analyzed (Participants) | 29
percentage of HbA1c | -2.82 (1.084)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 for Double-blind Group
Description: FPG was obtained at baseline and at Week 24. The model-adjusted change from baseline was calculated using mixed-effects repeated measures analysis.
Time Frame: Baseline, up to 24 weeks
Population: ITT population was used for the analysis. Subjects with a value at baseline and at week 24 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo
Number analyzed (Participants) | 142 | 145
mmol/L | -2.51 (0.174) | -1.16 (0.173)
Statistical Analysis 1: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -1.35, 95% CI 2-sided [-1.83 to -0.86]

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 for High Glycemic Group
Description: The change in FPG from baseline at Week 24 for High Glycemic Group was calculated by subtracting the mean FPG at baseline from the mean FPG at Week 24
Time Frame: Baseline, up to 24 weeks
Population: ITT population was used for the analysis. Subjects with a value at baseline and at week 24 were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | High Glycemic Group
Number analyzed (Participants) | 29
mmol/L | -4.98 (3.437)

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 24
Description: Changes from baseline at Week 24 in SBP for the double-blind group and high glycemic group
Time Frame: Baseline to week 24
Population: The ITT population was used for the analysis. Subjects with a value at baseline and at the specific visit were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo | High Glycemic Group
Number analyzed (Participants) | 143 | 145 | 29
mm Hg | -5.03 (0.993) | 2.04 (0.987) | -8.19 (14.882)
Statistical Analysis 1: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -7.07, 95% CI 2-sided [-9.83 to -4.32]

6. Secondary Outcome: Proportion of Subjects Achieving HbA1c < 7% Over Time for Double-blind Group
Description: The proportion of subjects who achieved HbA1c < 7% at 6, 12, 18 and 24 weeks were calculated based on the number of subjects with a value at each time point for each group. The model-adjusted proportion was calculated based on a logistic analysis using Generalized Estimating Equation (GEE) logistic regression that includes country, treatment, visit, treatment-by-visit interaction and the baseline HbA1c value as a fixed effect covariate. An unstructured correlation structure will be used, or autoregressive if the model with the unstructured structure does not converge.
Time Frame: Baseline, up to 24 weeks
Population: The number of subjects in the ITT population with a value at baseline and at the specified visit was included. Model-adjusted proportion (LS proportion) and 95% confidence interval were reported for Double-blind Treatment Group.
Measure: Least Squares Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo
Number analyzed (Participants) | 158 | 159
Proportion of subjects
  Week 6: number analyzed (Participants) | 152 | 152
  Week 6 | 0.14 [0.09 to 0.23] | 0.03 [0.01 to 0.07]
  Week 12: number analyzed (Participants) | 149 | 146
  Week 12 | 0.26 [0.18 to 0.38] | 0.06 [0.03 to 0.12]
  Week 18: number analyzed (Participants) | 143 | 144
  Week 18 | 0.26 [0.18 to 0.39] | 0.10 [0.06 to 0.18]
  Week 24: number analyzed (Participants) | 142 | 145
  Week 24 | 0.38 [0.26 to 0.55] | 0.10 [0.06 to 0.17]
Statistical Analysis 1: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Odds ratio at Week 6 was calculated as the odds ratio of bexagliflozin group over placebo group; Test type: Superiority; p = 0.0014, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.69, 95% CI 2-sided [1.70 to 12.95] — The odds ratios of bexagliflozin group over the placebo group at each visit will be estimated from LS means based on the model with the corresponding p-values and their two-sided 95% CIs presented
Statistical Analysis 2: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Odds ratio at Week 12 was calculated as the odds ratio of bexagliflozin group over placebo group; Test type: Superiority; p = 0.0001, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.18, 95% CI 2-sided [1.96 to 8.92] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Odds ratio at Week 18 was calculated as the odds ratio of bexagliflozin group over placebo group; Test type: Superiority; p = 0.0030, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.31 to 5.04] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Odds ratio at Week 24 was calculated as the odds ratio of bexagliflozin group over placebo group; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.88, 95% CI 2-sided [1.99 to 7.58] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Proportion of Subjects Achieving HbA1c < 7% Over Time for High Glycemic Group
Description: The proportion of subjects who achieved HbA1c < 7% at 6, 12, 18 and 24 weeks were calculated based on the number of subjects with a value at each time point for each group.
Time Frame: Baseline, up to 24 weeks
Population: The number of subjects in the ITT population with a value at baseline and at the specified visit was included. Proportion of subjects achieving HbA1c < 7% was reported for High Glycemic Group without a 95% confidence interval.
Measure: Number; unit: Proportion of subjects
Arm/Group | High Glycemic Group
Number analyzed (Participants) | 34
Proportion of subjects
  Week 6 | 0
  Week 12 | 0.065
  Week 18 | 0.097
  Week 24 | 0.138

8. Secondary Outcome: Change in Body Mass From Baseline to Week 24 in Subjects With a BMI ≥ 25 kg/m2 for Double-blind Group
Description: Changes in body mass from baseline to week 24 was calculated based on LS means for both bexagliflozin and placebo groups.
Time Frame: Baseline to week 24
Population: Subjects with a BMI >= 25 kg/m2 at baseline in the ITT population were included. The number of subjects with a value at baseline and at week 24 was analyzed. Model-adjusted mean change (LS Mean) and standard error (SE) were reported.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo
Number analyzed (Participants) | 119 | 124
kg | -3.60 (0.348) | -1.09 (0.336)
Statistical Analysis 1: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA analysis includes country, treatment, visit, treatment and baseline HbA1c value as fixed effect covariates; Difference of LS Means = -2.51, 95% CI 2-sided [-3.45 to -1.57]

9. Secondary Outcome: Change in Body Mass From Baseline to Week 24 in Subjects With a BMI ≥ 25 kg/m2 for High Glycemic Group
Description: The change in body mass from baseline at week 24 for High Glycemic group was calculated by subtracting the mean body mass at baseline from the mean body mass at week 24
Time Frame: Baseline to week 24
Population: Subjects with a BMI >= 25 kg/m2 at baseline in the ITT population were included. The number of subjects with a value at baseline and at week 24 was analyzed.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | High Glycemic Group
Number analyzed (Participants) | 28
kg | -1.40 (3.759)

10. Secondary Outcome: Change From Baseline in HbA1c Over Time in Double-blind Treatment Group
Description: The change from baseline in HbA1c at 6, 12, 18 and 24 weeks was calculated based on the number of subjects with a value at each time point for each group. The model-adjusted change from baseline was calculated based on a mixed-effects repeated measures analysis that includes country, treatment, visit, treatment-by-visit interaction and the baseline HbA1c value as a fixed effect covariate.
Time Frame: Baseline, up to 24 weeks
Population: The Number Analyzed only includes the number of subjects with a value at baseline and at the specific visit. Model-adjusted mean change (LS Mean) and standard error (SE) were reported for Double-blind Treatment Group.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo
Number analyzed (Participants) | 158 | 159
percentage of HbA1c
  Week 6: number analyzed (Participants) | 152 | 152
  Week 6 | -0.72 (0.065) | -0.16 (0.065)
  Week 12: number analyzed (Participants) | 149 | 146
  Week 12 | -0.97 (0.073) | -0.31 (0.073)
  Week 18: number analyzed (Participants) | 143 | 144
  Week 18 | -1.00 (0.072) | -0.51 (0.072)
  Week 24: number analyzed (Participants) | 142 | 145
  Week 24 | -1.09 (0.076) | -0.56 (0.075)
Statistical Analysis 1: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Model-adjusted change from baseline at week 6 was calculated as the difference in LS Mean between bexagliflozin group and placebo group; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.56, 95% CI 2-sided [-0.74 to -0.38]
Statistical Analysis 2: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Model-adjusted change from baseline at week 12 was calculated as the difference in LS Mean between bexagliflozin group and placebo group; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.66, 95% CI 2-sided [-0.86 to -0.46]
Statistical Analysis 3: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Model-adjusted change from baseline at week 18 was calculated as the difference in LS Mean between bexagliflozin group and placebo group; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.50, 95% CI 2-sided [-0.69 to -0.30]
Statistical Analysis 4: Comparison: Double-blind Group: Bexagliflozin 20 mg vs Double-blind Group: Placebo; Model-adjusted change from baseline at week 24 was calculated as the difference in LS Mean between bexagliflozin group and placebo group; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures — P-value is presented based on one-sided statistical tests using a 0.025 level of significance; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.53, 95% CI 2-sided [-0.74 to -0.32]

11. Secondary Outcome: Change in HbA1c Over Time Among Subjects Who Have Baseline HbA1c of > 10.5% and ≤ 12.0%
Description: The change from baseline in HbA1c at 6, 12, 18 and 24 weeks was calculated based on the number of subjects with a value at each time point in High Glycemic Group.
Time Frame: Baseline, up to 24 weeks
Population: The Number Analyzed only includes the number of subjects with a value at baseline and at the specific visit.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | High Glycemic Group
Number analyzed (Participants) | 34
percentage of HbA1c
  Week 6: number analyzed (Participants) | 28
  Week 6 | -1.72 (1.027)
  Week 12: number analyzed (Participants) | 31
  Week 12 | -2.45 (1.136)
  Week 18: number analyzed (Participants) | 31
  Week 18 | -2.62 (1.055)
  Week 24: number analyzed (Participants) | 29
  Week 24 | -2.82 (1.084)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Week -1 (run in period: Visit 2) to Week 26 (Follow up: Visit 8).
Arm/Group | Double-blind Group: Bexagliflozin 20 mg | Double-blind Group: Placebo | High Glycemic Group
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/159 | 0/34
Serious Adverse Events (participants affected / at risk) | 3/158 | 4/159 | 0/34
Other Adverse Events (participants affected / at risk) | 16/158 | 28/159 | 7/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Group: Bexagliflozin 20 mg (N=158) | Double-blind Group: Placebo (N=159) | High Glycemic Group (N=34)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Group: Bexagliflozin 20 mg (N=158) | Double-blind Group: Placebo (N=159) | High Glycemic Group (N=34)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 (3) | 10 (10) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (9) | 13 (13) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 5 (6) | 4 (4) | 3 (3)
Polyuria (Renal and urinary disorders) | 5 (7) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator does not have the right to publish trial results.

DOCUMENTS (2):
  • Study Protocol (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT03259789/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT03259789/SAP_001.pdf